CLINICAL TRIAL: NCT05250518
Title: Comparison of Argon Plasma Coagulation and Clip Closure for the Prophylaxis of Colorectal Post-polypectomy Bleeding After Hot Snare Polypectomy: a Multicenter, Randomized and Controlled Study
Brief Title: Argon Plasma Coagulation and Clip for the Prophylaxis of Post-polypectomy Bleeding After Hot Snare Polypectomy
Acronym: APC、HSP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, ChenMingkai, Professor, Renmin Hospital of Wuhan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WDRY2022-K018
Record Dates: First submitted 2022-02-18; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Post-polypectomy Bleeding; Colorectal Polyp
Keywords: hot snare polypectomy; argon plasma coagulation; clip closure
MeSH Terms: interventions — Argon Plasma Coagulation; Surgical Instruments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- the control group (No Intervention): The control group will receive no prophylaxis of post-procedure bleeding.
- APC group (Experimental): The APC group will receive prophylaxis of post-procedure bleeding with argon plasma coagulation.
  Interventions: Procedure: argon plasma coagulation
- Clip group (Experimental): The Clip group will receive prophylaxis of post-procedure bleeding with clip closure.
  Interventions: Procedure: clip closure

INTERVENTIONS:
Procedure: argon plasma coagulation — After hot snare polypectomy, participants will be randomized assigned to the APC group for argon plasma coagulation to prevent colorectal post-procedure bleeding.
  Arms: APC group
Procedure: clip closure — After hot snare polypectomy, participants will be randomized assigned to the Clip group for complete closure(spacing between adjacent clips < 1cm) to prevent colorectal post-procedure bleeding.
  Arms: Clip group

SUMMARY:
Discuss the efficacy and safety of argon plasma coagulation （APC）in comparison with clip closure for preventing colorectal post-procedure bleeding（PPB） after hot snare polypectomy（HSP）; analyze the risk factors and the cost-effectiveness of bleeding prophylaxis strategies with Decision Tree Analytical Method.

DETAILED DESCRIPTION:
This is a multicenter, randomized and controlled study. It aims to discuss the efficacy and safety of argon plasma coagulation（APC）in comparison with clip closure for preventing colorectal post-procedure bleeding（PPB） after hot snare polypectomy（HSP）, and analyze the risk factors and the cost-effectiveness of bleeding prophylaxis strategies with Decision Tree Analytical Method.

According to the prophylaxis measures, patients enrolled in this study will be randomized into the control group, APC group and Clip group. It will collect participants' data of baseline character, postoperative and follow-up. All statistical analyses will be performed by SPSS 26.0 and Tree Age Pro 2011.

Based on the previous studies, it is presumed that the rate of PPB for the control group, Clip group and APC group is 8%, 2% and 2%. Given two-side testing, an alpha of 0.05 and a power of 90%, allowing for a 5% dropout rate, the smallest sample size is 1287.

ELIGIBILITY:
Inclusion Criteria:

1. age>18 years
2. the diagnosis of colorectal polyps is clear（Paris Ip or Ⅰsp）
3. head diameter≥ 10 mm
4. HSP indications were met and no contraindications were found
5. patients (or the legal representative/guardian) with informed consent

Exclusion Criteria:

1. ASA Grade Ⅲ or above, or end-stage disease of major organs (such as malignancy, heart failure, chronic obstructive pulmonary disease, end-stage renal disease and so on)
2. coagulation dysfunction (INR ≥ 1.5, PLT < 50×10 ^9 / L)
3. use antiplatelet drugs within 7 days before the operation, anticoagulant drugs within 5 days, and/or blood products within 30 days after the operation
4. there were other lesions in the resection site of the included polyps affecting this study, or the intestinal preparation was insufficient
5. incomplete closure of clips (complete closure: spacing between adjacent clips < 1cm)
6. APC is used for polypectomy or intraoperative hemostasis, rather than preventing PPB
7. surgical treatment, vascular intervention, or blood products were used during the operation
8. use other methods to prevent PPB
9. the bleeding site was not confirmed by endoscopy
10. history of intestinal surgery
11. menstruation or pregnancy
12. not following medical advice
13. participated in other clinical trials and signed its informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1017 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
The rate of re-bleeding | 30 days after HSP
  the rate of re-bleeding within 30 days after operation

SECONDARY OUTCOMES:
Location of re-bleeding sites | 30 days after HSP
  the original polyps' location of re-bleeding sites: cecum, ascending colon, colonic hepatic flexure, transverse colon, colonic splenic flexure , descending colon, sigmoid colon, rectum
Other postoperative complications | 30 days after HSP
  Other postoperative complications (perforation, electrocoagulation syndrome after polypectomy, stenosis, etc.)
Expenses of prevention | the 1 day of discharge from medical centers
  Expenses of argon plasma coagulation and clips

CONTACTS AND LOCATIONS:
Overall Officials: Mingkai Chen, Ph.D & M.D, Study Director — Renmin Hospital of Wuhan University
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided
undecided